CLINICAL TRIAL: NCT05702125
Title: Chronic Pain After Cardiothoracic Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Ratna Farida Soenarto, Principal Investigator, Indonesia University
Other Study IDs: IndonesiaUAnes921
Record Dates: First submitted 2023-01-10; First posted 2023-01-27 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Chronic Pain; Thoracic; Chronic Pain Syndrome
Keywords: chronic pain; thoracotomy; sternotomy; cardiothoracic surgery
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective cohort study to estimate prevalence of chronic pain after cardiothoracic surgery

DETAILED DESCRIPTION:
This is a prospective cohort study of all patients undergo cardiothoracic elective surgery in Cipto Mangunkusumo Hospital using general anesthesia. Patients with emergency surgery, history of psychologic and neurologic disease which cannot reliably state their pain score, cannot communicate well, and disagree to follow the research will be exempted. The pain score will be recorded one week after surgery during walk-in consultation, followed by 3 months and 6 months after surgery via telecommunication.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergo elective sternotomy and/or thoracotomy using general anesthesia
* Patients agree to follow the study

Exclusion Criteria:

* Patients undergo emergency sternotomy or thoracotomy
* Patients with pyschological and neurological disorder, that it is not reliable to determine the pain intensity
* Patients who cannot communicate
* Patients disagree to follow the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergo elective sternotomy and/or thoracotomy using general anesthesia in Cipto Mangunkusumo hospital during January 2023 until March 2024
Sampling Method: Non-Probability Sample
Enrollment: 96 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | 1 week after surgery
  Pain score to assess pain intensity
Visual Analog Scale | 3 months after surgery
  Pain score to assess postoperative pain intensity
Visual Analog Scale | 6 months after surgery
  Pain score to assess postoperative pain intensity

CONTACTS AND LOCATIONS:
Overall Officials: Ratna F Soenarto, Consultant, Principal Investigator — Indonesia University